CLINICAL TRIAL: NCT04949230
Title: A Retrospective Study to Analyze Efficacy of COVID-19 Treatments
Brief Title: A Retrospective Study of COVID-19 Treatments
Status: Completed | Type: Observational
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Other Study IDs: PRG-051
Record Dates: First submitted 2021-06-29; First posted 2021-07-02 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Covid19; COVID-19 Pneumonia; COVID-19 Respiratory Infection; COVID-19 Acute Bronchitis; COVID-19 Acute Respiratory Distress Syndrome; COVID-19 Lower Respiratory Infection; SARS-CoV2 Infection; SARS-CoV-2 Acute Respiratory Disease
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Patients: Subjects who have recovered from COVID-19
  Interventions: Other: No Intervention Used

INTERVENTIONS:
Other: No Intervention Used — There is no intervention in this study

SUMMARY:
Surveys administered to subjects who have recovered from COVID-19 to assess how effective their treatment was.

DETAILED DESCRIPTION:
Subjects who have recovered from COVID-19 will answer questions regarding the severity of their illness, symptoms experienced, what treatment they received, and how long they were ill.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, demonstrating that the patient understands the procedures required for the study and the purpose of the study
2. Male or female of 18 years of age or older
3. Diagnosis of COVID-19 infection by RT- PCR
4. Recovery from COVID-19

Exclusion Criteria:

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Refusal to sign informed consent form
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Survey Response | One hour
  Answers given by subjects on their recovery from COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Study Director — ProgenaBiome
Locations (1):
- Ginger Aurella, Ventura, California, United States